CLINICAL TRIAL: NCT00389987
Title: A Prospective, Multicenter, Double-Blind With In-House Blinding, Randomized, Comparative Study to Evaluate the Efficacy, Safety, and Tolerability of Ertapenem Sodium Versus Piperacillin/Tazobactam in the Treatment of Complicated Intra-Abdominal Infections in Hospitalized Adults
Brief Title: Ertapenem Sodium vs. Piperacillin/Tazobactam in the Treatment of Complicated Intra-Abdominal Infections (0826-037)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0826-037; 2006_538
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Complicated Intra-Abdominal Infections
MeSH Terms: interventions — Ertapenem; Duration of Therapy; Tazobactam

INTERVENTIONS:
Drug: MK0826, /Duration of Treatment : 8 Weeks
Drug: Comparator : piperacillin sodium (+) tazobactam sodium /Duration of Treatment : 8 Weeks

SUMMARY:
This study is designed to compare the efficacy of ertapenem and piperacillin/tazobactam with respect to the clinical response in baseline microbiologically evaluable patients; and to evaluate the tolerability and safety of ertapenem compared to piperacillin/tazobactam.

DETAILED DESCRIPTION:
Original label approved November 2001

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients (greater or equal to 18 years of age)
* Intraoperative/Postoperative Enrollment: Upon visual confirmation of an intra-abdominal infection.
* Preoperative Enrollment: Patients may be enrolled preoperatively if they meet certain criteria

Exclusion Criteria:

* Failure to meet all inclusion criteria.
* Patients who are considered unlikely to survive the 6-8 week study period.
* Pregnant or nursing women, or fertile women not practicing adequate methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-09; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
In microbiologically evaluable patients, ertapenem will be at least as effective as piperacillin/tazobactam at the 2-weeks post-treatment Early Follow-up Assessment. | 2-weeks post-treatment

SECONDARY OUTCOMES:
In microbiologically evaluable patients, ertapenem will be at least as effective as piperacillin/tazobactam at the 4-6 weeks post-treatment Late Follow-up Assessment. | 4-6 Weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Namias N, Solomkin JS, Jensen EH, Tomassini JE, Abramson MA. Randomized, multicenter, double-blind study of efficacy, safety, and tolerability of intravenous ertapenem versus piperacillin/tazobactam in treatment of complicated intra-abdominal infections in hospitalized adults. Surg Infect (Larchmt). 2007 Feb;8(1):15-28. doi: 10.1089/sur.2006.030. PMID 17381394
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html